CLINICAL TRIAL: NCT04646564
Title: Systemic Therapy With or Without Local Radiotherapy for Extracranial Oligometastatic Breast Cancer
Brief Title: Radiotherapy for Extracranial Oligometastatic Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Wuhan University (Other); China-Japan Union Hospital, Jilin University (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); West China Hospital (Other); Shanxi Province Cancer Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Shu lian Wang, Clinical professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2493
Record Dates: First submitted 2020-11-10; First posted 2020-11-30 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer Metastatic
Keywords: breast neoplasm; oligometastases; radiotherapy; stereotactic ablative radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (Active Comparator): standard of care
  Interventions: Drug: standard of care
- study arm (Experimental): radiotherapy + standard of care
  Interventions: Drug: standard of care; Radiation: radiotherapy + standard of care

INTERVENTIONS:
Drug: standard of care — patients receive appropriate therapy at the discretion of the treating oncologist, i.e. systemic therapy according to molecular subtypes, including chemotherapy, endocrine therapy, targeted therapy, or immunotherapy.
Radiation: radiotherapy + standard of care — Patients receive radiotherapy to all known metastases. SBRT technique is preferred, especially for metastases in bone, lung and liver. Conventional RT can be used when SBRT is not appropriate, such as metastasis in mediastinal or contralateral supraclavicular nodal regions. Total doses of 30Gy to 50Gy in 5 fractions for SBRT are recommended depending on the tolerance of adjacent normal tissue. Total dose of 60Gy in 25 fractions is recommended for conventional RT.
  Patients can receive systemic therapy concurrently with RT at the discretion of treating radiation oncologist. After completion of SBRT to all sites of known metastatic disease, patients will continue standard of care therapy per the treating oncologist.
  Arms: study arm

SUMMARY:
More and more evidence suggests that local radiotherapy can improve the outcomes for patients with oligometastatic disease. The purpose of this study is to assess the impact of radiotherapy, compared with standard systemic therapy alone, on survival, local control and toxicities in patients with extracranial oligometastatic breast cancer. Eligible patients are randomized in a 1:2 ratio between the control arm (standard systemic therapy), and the WLRT arm (standard systemic therapy + radiotherapy). Randomization will be stratified by three factors: visceral metastasis (yes vs.no), number of metastases(≤2 vs. >2), hormone receptor(positive vs. negative). SBRT technique is preferred. During and after radiotherapy, the patients are followed and the efficacy and toxicities of radiotherapy are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* ECOG performance status 0-2.
* Newly-diagnosed or metachronous extracranial oligometastatic diseases confirmed by pathology or imaging, with or without locoregional disease (biopsy of metastasis is preferred).
* Total number of locoregional and metastatic lesions of 1-5 , the maximum diameter of lesions ≤5 cm and at least one lesion could be evaluated by RECIST1.1.
* Have received or plan to receive systemic therapy.
* All lesions could be safely treated by radiotherapy.
* Life expectancy > 6 months.
* Have adequate organ function.

Exclusion Criteria:

* Have metastases in the central nervous system.
* have indications for palliative radiotherapy to reduce symptoms, such as pain, bleeding, obstruction, and pending fractures caused by the tumor.
* Have moderate/severe liver dysfunction (Child Pugh B or C) from liver metastases, .
* Malignant pleural effusion
* Unable to tolerate radiotherapy due to serious comorbidity
* Have received prior radiotherapy for target area
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  Time from randomization to disease progression at any site or death.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Time from randomization to death from any cause.
Local control rate | 2 years
  Incidence of tumor control within RT fields during follow up.
Incidence of toxicities | 2 years
  Incidence of acute and late toxicities from treatment graded according to radiation therapy oncology group (RTOG) radiation injury criteria and National Cancer Institute CTCAE version 4.0
Quality of Life measured by the Functional Assessment of Cancer Therapy- General (FACT-G) | 2 years
  Assessment of quality of life scores by FACT-G
Translational exploration | 2 years
  Assessment of circulating tumor cells (CTCs), ctDNA, as prognostic and predictive markers of survival, and for early detection of progression.
Proportion of acceptable SBRT completion | 2 years
  Proportion of patients who completed SBRT with acceptable dose prescriptions

CONTACTS AND LOCATIONS:
Overall Officials: Shu-lian Wang, M.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Wei-Fang Yang, Taizhou, Zhejiang